CLINICAL TRIAL: NCT02436993
Title: A Phase II Study of Breast Cancer Treatment Using Weekly Carboplatin + Paclitaxel With Pertuzumab + Trastuzumab (HER2+) or Bevacizumab (HER2-) in the Neoadjuvant Setting
Brief Title: Phase II Breast Ca Carboplatin + Paclitaxel With Pertuzumab + Trastuzumab or Bevacizumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Rita Sanghvi, Mehta, HS Clinical Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20151888; UCI 14-67 (Other: CFCCC)
Record Dates: First submitted 2015-04-20; First posted 2015-05-07 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Breast Carcinoma
Keywords: Neoadjuvant Treatment; Carboplatin; Paclitaxel; Pertuzumab; Trastuzumab; Bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin+Paclitaxel+Bevacizumab (HER2-) (Experimental): Carboplatin weekly 12 doses Paclitaxel weekly 12 doses Bevacizumab every other week, 5 doses
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab
- Carboplatin+Paclitaxel+Trastuzumab+Pertuzumab (HER2+) (Experimental): Carboplatin weekly 12 doses Paclitaxel weekly 12 doses Trastuzumab weekly 12 doses Pertuzumab every 3 weeks, 4 doses
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Carboplatin — Area Under the Curve (AUC) 2 IV over 60 minutes weekly for 12 doses
  Other Names: Paraplatin
Drug: Paclitaxel — 80 mg/m^2 IV over 1-3 hours weekly for 12 doses
  Other Names: Taxol
Drug: Bevacizumab — 10mg/kg IV over 90 or 60 or 30 minutes every other week for 5 doses
  Other Names: Avastin
  Arms: Carboplatin+Paclitaxel+Bevacizumab (HER2-)
Drug: Trastuzumab — 4mg/kg induction, followed by weekly 2mg/kg IV-induction over 90 minutes, then weekly over 30-60 minutes for 12 doses
  Other Names: Herceptin
  Arms: Carboplatin+Paclitaxel+Trastuzumab+Pertuzumab (HER2+)
Drug: Pertuzumab — 840mg induction, followed by 420mg every 3 weeks IV-induction over 60 minutes, then every 3 weeks over 30-60 minutes for 4 doses
  Other Names: Perjeta
  Arms: Carboplatin+Paclitaxel+Trastuzumab+Pertuzumab (HER2+)

SUMMARY:
The purpose of this phase II is to study the efficacy and toxicity of carboplatin and paclitaxel with pertuzumab and trastuzumab in HER2 positive and carboplatin and paclitaxel with bevacizumab in HER2 negative in the neoadjuvant setting for the treatment of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES The study component is to evaluate the treatment response and toxicity of the protocol.

Objectives for treatment study component:

1.1 To estimate 2-year progression-free survival in patients with breast cancer with tumor more than 1 cm and/or with clinically detected lymph node treated with neoadjuvant weekly Carboplatin and Paclitaxel combined with Trastuzumab + Pertuzumab in HER2-positive disease or with Bevacizumab in HER2-negative disease.

1.2 To measure the microscopic complete pathological response (pCR) rates defined as ypT0 or ypTis tumors in patients treated with this regimen in the neoadjuvant setting.

1.3 To assess complete clinical response (cCR) rates after treatment by physical exam and imaging tests (ultrasonography, mammography, or magnetic resonance imaging) clinical objective response rate (by Response Evaluation Criteria In Solid Tumors (RECIST)) 1.4 To determine the toxicity of this regimen. 1.5 To determine treatment adherence and delivered dose intensity of this regimen.

1.6 To assess the correlation between pCR and cCR. 1.7 To determine the rate of breast conservation following neoadjuvant therapy. 1.8 Determine treatment efficacy according to subgroups defined according to stage and receptor status.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven unilateral or bilateral primary breast carcinoma. (In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.)
2. Tumor size is clinically at least 1 cm in greatest diameter (palpable or by imaging) and/or with involved lymph node. In case of inflammatory disease, the extent of inflammation may be the measurable lesion.
3. Documentation of inflammatory breast cancer
4. Woman age > or = 18
5. Performance status of 0-2 by Eastern Cooperative Oncology Group (ECOG) criteria
6. Known HER2 status
7. Normal cardiac function must be documented within 90 days prior to registration either via an ECHO or MUGA or per physician's review of symptoms and medical history. If an ECHO is performed as standard of care, the ejection fraction must be above the normal limit of the institution.. If not available in the medical chart, the ECHOs or MUGAs are not required to be repeated for research purposes.

   a. Date of Echo or multigated acquisition (MUGA) (within 90 days) if performed
8. Staging work-up prior to registration

   1. Date of physical examination (within 90 days)
   2. Date of bilateral mammogram (within 90 days)
   3. Date of breast ultrasound (within 90 days)
   4. Date of MRI breast (within 30 days)
   5. Chest X-ray or CT- Chest or CT/PET Scan that includes the Chest may be done at physician's discretion (within 90 days). If not available in the medical chart, the Chest X-ray or CT- Chest or CT/PET Scan that includes the Chest is not required to be repeated for research purposes.
   6. Other tests as clinically indicated
9. Laboratory requirements:

   1. Hematology:

      * Absolute Neutrophil Count (ANC) ≥ 1,500/μl
      * Platelets ≥ 100,000/μl
   2. Hepatic Function

      * Total Bilirubin <1x upper limit of normal (ULN)
      * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x ULN
   3. Renal Function

      - Creatinine <1.5x ULN
   4. Proteinuria

      - Random urine total protein <100mg/dL. Urine Protein Creatinine (UPC) ratio <2g
   5. Negative pregnancy test for women of childbearing potential within 14 days prior to registration.
10. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

    Exclusion Criteria:
11. Evidence of distant metastasis. If radiographic suspicion of distant metastatic site, a negative biopsy must be available in the medical record. If not available in the medical record, the subject may be included and a confirmatory biopsy is not required to be performed for research purposes.
12. Known or suspected congestive heart failure, angina pectoris requiring antianginal medication, or other clinically significant cardiac condition.
13. Pregnant or nursing women may not participate due to the possibility of harm to fetus or nursing infants from this treatment regimen. Women of childbearing potential may not participate unless they have agreed to use an adequate contraceptive method throughout study treatment and for one month after completion of treatment.
14. Male patients
15. Pre-existing peripheral neuropathy of severity grade ≥ 2 (limiting instrumental activities of daily living).
16. Incomplete wound healing.
17. Active and significant bleeding
18. Known allergy, hypersensitivity or prior infusion reaction to one or more of the therapies incorporated into this treatment protocol.
19. Bone marrow depression or hematologic parameters in the range that would increase the risk for severe bleeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04; Primary Completion 2023-11 (Actual); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival in patients treated with weekly carboplatin and paclitaxel combined with either trastuzumab and pertuzumab for HER2-positive patients or bevacizumab for HER2-negative patients in the neoadjuvant setting | 2 years
  Progression of disease-A new lesion or a greater than or equal to 25% increase in the product of the largest perpendicular diameters of any one lesion on clinical exam or by U/S or MRI Survival-from date of registration to date of death

SECONDARY OUTCOMES:
Clinical complete response rates | 2 years
  Clinical complete response (cCR)-Normal breast on physical exam. No mass, no thickening, no erythema, no peau d'orange
Pathologic complete response rates | 2 years
  Pathologic complete response (pCR)-No histologic evidence of microscopic invasive tumor at the primary tumor site in the surgical specimen (ypT0 or DCis)
Number of toxicities in Carboplatin+Paclitaxel+Bevacizumab (HER2) arm | Up to 42 days after discontinued treatment
  This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 for toxicity and Adverse Event reporting.
Number of toxicities in Carboplatin+Paclitaxel+Trastuzumab+Pertuzumab (HER2+) | Up to 42 days after discontinued treatment
  This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 for toxicity and Adverse Event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California, United States